CLINICAL TRIAL: NCT04359420
Title: What Are the Benefits and Harms of Risk Stratified Screening as Part of the NHS Breast Screening Programme: Study Protocol for a Multi-site Non-randomised Comparison of BC-Predict Versus Usual Screening
Brief Title: What Are the Benefits and Harms of Risk Stratified Screening in the NHS Breast Screening Programme: Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Breast Cancer Now (Other); Prevent Breast Cancer (Unknown); Queen Mary University of London (Other); University of Nottingham (Other); Manchester University NHS Foundation Trust (Other Government); East Lancashire Hospitals NHS Trust (Other); East Cheshire NHS Trust (Unknown); NHS Breast Screening Programme (Unknown); The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David French, Prof David French, University of Manchester
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RP-PG-1214-20016
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; Screening; risk stratification; high risk; psychological impact; early detection; mammographic density; chemoprevention; Tyrer-Cuzick; anxiety
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A non-randomised fully counterbalanced study design will be used, to include equal numbers of participants from all sites who will be offered NHS-BSP and BC-Predict. Specifically, in the initial 8-month time period, women eligible for breast screening in three screening sites will be offered BC-Predict, whilst women in two screening sites are offered usual NHS-BSP. In the following 8-month time period the study sites switch to offer the other intervention (NHS-BSP rather than BC-Predict; and vice versa). This will allow estimates of effect to be obtained from both within-sample and between-sample analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BC-Predict (Experimental): Women will be sent an invitation letter one to two days after their breast screening invitation letter, directing prospective participants to the online risk assessment platform. Once participants have consented to the study online, they will be directed to the BC-Predict risk assessment questionnaire. Assessment of the online questionnaire during the pilot phase estimated that most women would be able to complete this within 30 minutes.
  Women who complete the questionnaire will receive 10-year breast cancer risk estimates once they have screened negative for breast cancer, based on the Tyrer-Cuzick model, incorporating mammographic density, and for some women, SNPs (single nucleotide polymorphisms). Women who are identified as being at "high" (>8%) or "moderate" (5% and <8%) 10-year risk will be offered a consultation to discuss prevention options including prescription of chemoprevention drugs and/ or more frequent mammography as part of the NHS Breast Screening Programme.
  Interventions: Other: BC-Predict
- NHS-Breast Screening Programme (Active Comparator): Usual care in the NHS Breast Screening Programme, which involves mammography every 3 years for the majority of women
  Interventions: Other: NHS Breast Screening Programme

INTERVENTIONS:
Other: BC-Predict — BC-Predict is an automated system for offering an assessment of breast cancer risk to women when they receive their NHS Breast Screening Programme invitation, and generating letters to feedback this risk to women and relevant healthcare professionals. Women at higher risk are offered chemoprevention drugs and additional mammography
  Other Names: risk stratified screening
  Arms: BC-Predict
Other: NHS Breast Screening Programme — usual care from NHS Breast Screening Programme, consisting of mammography every three years for most women.
  Arms: NHS-Breast Screening Programme

SUMMARY:
This study aims to identify key benefits and harms of integrating risk stratification (the BC-Predict intervention) into the NHS Breast Screening Programme. A non-randomised fully counterbalanced study design will be used, whereby women from screening sites will be offered usual NHS Breast Screening Programme or BC-Predict for an eight month period, followed by a cross-over point where women at each site will be offered the other invention during an eight month period.

DETAILED DESCRIPTION:
In principle, risk-stratification as a routine part of the NHS breast screening programme (NHS-BSP) should produce a better balance of benefits and harms. The main benefit is the offer of NICE (National Institute of Health and Care Excellence) approved more frequent screening and/ or chemoprevention to be realised for women who are at increased risk, but are unaware of this. The invesigators have developed BC-Predict, which is offered to women when invited to NHS-BSP and collects information on risk factors (self-reported information on family history and hormone-related factors, mammographic density and in a sub-sample, Single Nucleotide Polymorphisms). BC-Predict then produces risk feedback letters, and invites women at moderate or high risk to have discussion of prevention and early detection options at Family History, Risk and Prevention Clinics. Key objectives of the present research are to quantify important potential benefits and harms, and to identify the key drivers of the relative cost-effectiveness of embedding BC-Predict into NHS-BSP.

A non-randomised fully counterbalanced study design will be used, to include equal numbers of participants from five screening sites who will be offered NHS-BSP and BC-Predict. Specifically, in the initial 8-month time period, women eligible for NHS-BSP in three screening sites will be offered BC-Predict, whilst women in two screening sites are offered usual NHS-BSP. In the following 8-month time period the study sites switch their offers. In total 16000 women will be invited to BC-Predict, and compared with 16000 women offered standard NHS-BSP. Key potential benefits including uptake of BC-Predict, risk consultations, chemoprevention and additional screening will be obtained from NHS-BSP and Family History, Risk and Prevention Clinic records for both groups. Key potential harms such as increased anxiety will be obtained via self-report questionnaires. Health economic analyses will identify the key uncertainties underpinning the relative cost-effectiveness of embedding BC-Predict into NHS-BSP.

ELIGIBILITY:
Inclusion Criteria:

* born biologically female,
* invited for either (a) first breast screening appointment (any age) or: (b) aged 57-63 years (only at East Cheshire and East Lancashire breast screening programmes),
* able to provide informed consent and complete a risk assessment questionnaire.

Exclusion Criteria:

* previously has had breast cancer,
* has had bilateral mastectomy, or
* has previously participated in the related PROCAS (Predicting Risk Of Cancer At Screening) study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32298 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Prescription of chemoprevention. | 6 months after screening appointment
  Frequency of women taking up initial prescription of chemoprevention drugs (anastrozole/tamoxifen/raloxifene) from Family History, Risk and Prevention Clinic
  Data will be collected on each of the following aspects of this: (a) participant agrees/disagrees in clinic to take chemoprevention, (b) chemoprevention not appropriate, (c) chemoprevention appropriate but prescription not filled, (d) chemoprevention appropriate and prescription filled.

SECONDARY OUTCOMES:
Screening attendance at first offered screening episode | attendance within 6 weeks of first specific appointment offered
  Attendance at NHS Breast Screening Programme appointment
Screening attendance within 180 days | within 180 days first appointment offered
  Attendance at NHS Breast Screening Programme appointment
number of recalls | within 6 months of first appointment offered
  number of recalls from NHS Breast Screening programme: (a) technical recalls, (b) for assessment, (c) routine recalls
Number of breast cancer diagnoses | within 6 months of first appointment offered
  Number of breast cancers diagnosed
Uptake of consultation at Family History, Risk and Prevention clinics | within 6 months of first appointment offered
  Family History, Risk and Prevention clinic attendance, to discuss possibly measures to reduce breast cancer risk
Enrolment for more frequent screening | within 6 months of first appointment offered
  Uptake of more frequent screening (e.g. yearly) from NHS Breast Screening programme
State anxiety | at 6 months of first appointment offered, controlling for baseline values
  Measured using STAI (Spielberger State Anxiety Inventory) short form. Range 6 to 24. Higher scores indicate higher anxiety.
Cancer worry | at 6 months of first appointment offered, controlling for baseline values
  Measured using Lerman Cancer Worry Scale. Range 6 to 24. Higher scores indicate higher cancer worry.
Informed choices to attend screening or not | at 6 months of first appointment offered, controlling for baseline values
  Informed choices regarding screening will be estimated from attitudes to screening at baseline, knowledge and screening attendance, using a standard approach reported by Marteau, Dormandy & Michie

OTHER OUTCOMES:
Cost consequences | at 6 months of first appointment offered
  cost consequences analysis to understand the short-term relative impact of the risk feedback intervention (BC-Predict) based on health status (EQ-5D5L), capability (ICECAP-A); and proportion of women starting chemoprevention.
Variation in uptake of services offered examined by deciles of index of multiple deprivation (as assessed using residential postcode) | at 6 months of first appointment
  The investigators will examine variations in proportion of people offered services (i.e. uptake of NHS Breast Screening programme and BC-Predict), between groups defined by deciles of Indices of Multiple Deprivation (derived from residential postcode). This will assess any potential exacerbation of health inequalities brought about by BC-Predict.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Evans, MD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be shared in anonymised format with bone fide researchers, once main outcomes from the study have been published.

REFERENCES:
- [Derived] Gareth Evans D, McWilliams L, Astley S, Brentnall AR, Cuzick J, Dobrashian R, Duffy SW, Gorman LS, Harkness EF, Harrison F, Harvie M, Jerrison A, Machin M, Maxwell AJ, Howell SJ, Wright SJ, Payne K, Qureshi N, Ruane H, Southworth J, Fox L, Bowers S, Hutchinson G, Thorpe E, Ulph F, Woof V, Howell A, French DP. Quantifying the effects of risk-stratified breast cancer screening when delivered in real time as routine practice versus usual screening: the BC-Predict non-randomised controlled study (NCT04359420). Br J Cancer. 2023 Jun;128(11):2063-2071. doi: 10.1038/s41416-023-02250-w. Epub 2023 Apr 1. PMID 37005486
- [Derived] Pegington M, Harvie M, Harkness EF, Brentnall A, Malcomson L, Southworth J, Fox J, Howell A, Cuzick J, Evans DG. Obesity at age 20 and weight gain during adulthood increase risk of total and premature all-cause mortality: findings from women attending breast screening in Manchester. BMC Womens Health. 2023 Jan 13;23(1):17. doi: 10.1186/s12905-023-02162-0. PMID 36635680
- [Derived] French DP, Astley S, Brentnall AR, Cuzick J, Dobrashian R, Duffy SW, Gorman LS, Harkness EF, Harrison F, Harvie M, Howell A, Jerrison A, Machin M, Maxwell AJ, McWilliams L, Payne K, Qureshi N, Ruane H, Sampson S, Stavrinos P, Thorpe E, Ulph F, van Staa T, Woof V, Evans DG. What are the benefits and harms of risk stratified screening as part of the NHS breast screening Programme? Study protocol for a multi-site non-randomised comparison of BC-predict versus usual screening (NCT04359420). BMC Cancer. 2020 Jun 18;20(1):570. doi: 10.1186/s12885-020-07054-2. PMID 32552763